CLINICAL TRIAL: NCT05144594
Title: Assessment of Direct Medical Costs Associated With Making a Negative Diagnosis of IBS.
Brief Title: Direct Medical Costs Associated With Negative Diagnosis of IBS.
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Region Örebro County (Other)
Responsible Party: Sponsor
Other Study IDs: 277075
Record Dates: First submitted 2021-11-22; First posted 2021-12-03 (Actual); Last update posted 2021-12-03 (Actual); Status verified 2021-11

CONDITIONS: Irritable Bowel Syndrome
Keywords: Irritable bowel syndrome; Rome IV; Functional gastrointestinal disorders
MeSH Terms: conditions — Irritable Bowel Syndrome; Gastrointestinal Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients diagnosed with IBS: Patients diagnosed with IBS within primary care in Region Örebro County between 2013-2017, identified by ICD-code K.58.

SUMMARY:
The purpose of this study is to calculate the unnecessary costs that are associated with a negative IBS diagnosis.

DETAILED DESCRIPTION:
In Örebro Region there are 29 public general health centers. Approximately 300.000 inhabitants are listed within these health centers. Approximately 150 doctors are currently working within the primary health care of Örebro Region. The electronic patient register in Örebro Region allows to search for the International Statistical Classification of Diseases (ICD-10) for IBS (K58.9 and K58.0) This allows retrospective research regarding diagnosis of IBS.

A study planned ahead of this study by the same research group will focus on adherence to guidelines of making a positive diagnosis of IBS. This data will be used for this study as well.

Data will be collected retrospectively over the period 2013-2017 using the the electronic patient register in Örebro Region. Patients diagnosed with IBS will be identified by ICD-code K.58. By evaluating their patient register it will be determined how the GP has made the IBS diagnosis. Patients will fall into three categories: those who received a positive IBS diagnosis using the Rome criteria, those who received a negative IBS diagnosis and those whose patient record is lacking sufficient information.

A detailed analysis of the collected data will focus on the proportion of patients who received a negative diagnosis. We will only include patients with age >40 years without "red flags", since in these patients additional diagnostics are seldom warranted and generally not useful. Red flags are, for example, blood in the stool, fever, anemia or involuntary weight loss. In patients over 40 years, certain additional diagnostics may be important. For example, changes in bowel habits may be caused by colorectal cancer and for this reason these patients are routinely referred for a colonoscopy according to the guidelines for the "standardized care chain".

For each patient, data regarding the used diagnostic tools will be collected and at the end the costs of these diagnostic tools will be calculated. If a patient is referred to a specialist, the costs for the associated diagnostics will be calculated as well.

The results of the diagnostic tests will be evaluated as well, in order to confirm that these tests were not indicated, as one may expect. If a patient was referred to a specialist, the costs for the associated diagnostics will be calculated as well. Diagnostic tools include gastroscopy, colonoscopy, abdominal ultrasound, vaginal ultrasound, abdominal x-ray and abdominal MRI. Laboratory testing includes liver tests, tests for lactose intolerance, stool samples, food allergy tests and autoimmune serology.

The two groups (positive vs negative diagnosis) will be compared regarding the costs of diagnostic tools and laboratory testing, in order to establish the total amount of costs that are associated with making a negative IBS diagnosis.

Descriptive statistical analysis of the economic costs for IBS patients receiving a positive diagnosis will be compared to those receiving a negative diagnosis. The total cost of all diagnostic procedures will be analyzed, as well as various cost components. A separate analysis will be performed to confirm the expected negative results of the additional diagnostic tests, associated with a negative IBS diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients (both sexes) who were diagnosed with IBS according to ICD-10 within primary care of Region Örebro County 2013-2017.

Exclusion Criteria:

* Patients < 18 years or > 65 years

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with IBS within primary care of Region Örebro County 2013-2017.
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2021-11-29 (Estimated); Primary Completion 2024-05-31 (Estimated); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
Direct medical costs of diagnostic tools associated with a negative diagnosis of IBS. | 2013-2017
  Unnecessary costs of diagnostic tools, e.g. endoscopy and radiology in SEK that are associated with a negative IBS diagnosis
Direct medical costs of laboratory tests associated with a negative diagnosis of IBS. | 2013-2017
  Unnecessary costs of laboratory tests, e.g. liver tests, tests for lactose intolerance, stool samples, food allergy tests and autoimmune serology, in SEK that are associated with a negative IBS diagnosis
Direct medical costs of referrals to specialists associated with a negative diagnosis of IBS. | 2013-2017
  Unncessary costs of referrals to specialist care. If a patient was referred to a specialist, the costs for the associated diagnostics will be calculated as well.

CONTACTS AND LOCATIONS:
Overall Officials: Michiel van Nieuwenhoven, M.D. Ph.D., Principal Investigator — Region Örebro County

IPD SHARING:
Plan to Share IPD: Undecided